CLINICAL TRIAL: NCT05426655
Title: Effects of a Self-management Program for Temporomandibular Myalgia in Subjects With Fibromyalgia: a Single Arm Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Edgar Ferrandez Gomez (Other)
Responsible Party: Sponsor-Investigator, Jose Edgar Ferrandez Gomez, Principal Investigator, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFG012022
Record Dates: First submitted 2022-06-13; First posted 2022-06-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Temporomandibular Disorder; Fibromyalgia; Self Management
Keywords: self-management; self-care; pain neuroscience education; temporomandibular disorder; fibromyalgia
MeSH Terms: conditions — Temporomandibular Joint Disorders; Fibromyalgia | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: Analytical, prospective experimental study: uncontrolled clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self management (Experimental): Intervention group: education in pain neuroscience + self-massage + exercises + advice and recommendations.
  Interventions: Other: Self management

INTERVENTIONS:
Other: Self management — The program will consist of 3 sessions in which everything related to pain and its management will be explained. In a first workshop, a first educational session on the neurophysiology of pain will be given by means of a Power Point presentation. In a second workshop, a tool will be used to locate those factors that can improve/worse the pain, physical documentation will be delivered with instructions for performing a self-massage and exercises of the temporomandibular region as well as advice and recommendations to manage different situations that may appear on a daily basis and on Lifestyle. A meditation session will also be held. In the third and last workshop, the game "the painometer" will be played and a meditation session will be held.

SUMMARY:
Fibromyalgia is one of the most prevalent chronic widespread pain entities today. One of the most common problems in patients with fibromyalgia are alterations of the temporomandibular region, present in approximately 80% of the subjects, being, in turn, alterations of muscular origin the most common with a prevalence of 84%. One of the most promising therapeutic strategies is one that leads to self-management by the patient. The main objective of this study is to analyze the effect of a self-management program for myalgia in the temporomandibular region in subjects with fibromyalgia. For this, an experimental study of the uncontrolled Clinical Trial type will be carried out. Participants must be over 18 years of age, have a diagnosis of fibromyalgia and have myalgia or myofascial pain syndrome in the temporomandibular region. Demographic data, mandibular function, pain level, quality of life related to oral health, kinesiophobia, anxiety and depression, sleep, patient oral habits, catastrophizing, knowledge about pain, central sensitization, self-efficacy, coping with pain patient expectations, and patient satisfaction with the treatment received. An initial data collection will be carried out. The intervention will be carried out in 3 online sessions in which different pain processes will be explained, mandibular mobility exercises, masticatory muscle self-massage, as well as recommendations and advice on its pathology. Data will be collected again 4 weeks after the end of the program and at months 6 and 12. The appearance of adverse effects linked to the therapeutic program is not contemplated.

DETAILED DESCRIPTION:
Study design Analytical, prospective experimental study: uncontrolled clinical trial.

Population and study sample The study sample will be made up of subjects diagnosed with fibromyalgia who present with local myalgia, myofascial pain or referred myofascial pain in the temporomandibular region, according to the diagnostic criteria (DC/TMD). The subjects will be recruited after the mandatory acceptance and authorization by the corresponding bodies, during a recruitment period of approximately eight weeks, through different associations of fibromyalgia patients.

Intervention In a first visit, demographic data will be recorded and an examination will be performed to assess the presence of local myalgia, myofascial pain or referred myofascial pain in the temporomandibular region, according to the diagnostic criteria (DC/TMD). You will also be given, to read and sign, the informed consent for participation in the study, as well as the data protection document. After this visit, the defined eligibility criteria (inclusion and exclusion) will be applied.

In a second visit, a preliminary assessment will be carried out that will consist of mandibular function, pain level, quality of life related to oral health, kinesiophobia, anxiety and depression, sleep, patient oral habits, catastrophizing, knowledge about pain, central sensitization, self-efficacy, coping with pain patient expectations, and patient satisfaction with the treatment received.

One week later, the intervention program will begin. The program will consist of 3 online sessions (visits 3, 4 and 5) in which everything related to pain and its management will be explained. In a first workshop, a first educational session on the neurophysiology of pain will be given by means of a Power point presentation. In a second workshop, a tool will be used to locate those factors that can improve/worse the pain, physical documentation will be delivered with instructions for performing a self-massage and exercises of the temporomandibular region as well as advice and recommendations to manage different situations that may appear on a daily basis and on Lifestyle. A meditation session will also be held. In the third and last workshop, the game "the painometer" will be played and a meditation session will be held.

On a sixth visit, 4 weeks after the end of the program, a new measurement and assessment will be taken. This measurement will be very similar to the one performed on the second visit, except for 1 variable: the patient's expectations will not be recorded, and the patient's satisfaction with the treatment received will be recorded. The objective will be to record the changes produced after the application of the treatment program.

On a seventh visit, at 6 months (medium-term follow-up), all the measurements and assessments made on the sixth visit will be repeated, with the aim of recording their status after six months.

At an eighth visit, at 12 months (long-term follow-up), all the measurements and assessments made at the seventh visit will be repeated, with the aim of recording their status after twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old.
* Subjects diagnosed with fibromyalgia.
* Orofacial pain of at least 3 months of evolution (considered chronic, according to IASP).
* Presence of myalgia, local myalgia, myofascial pain or referred myofascial pain in the temporomandibular region (according to DC/TMD).

Exclusion Criteria:

* Internal temporal-romandibular joint disorder with anterior disc displacement, joint pathology (arthritis), facial paralysis (active), mandibular fracture (active), infectious-inflammatory picture of odontogenic origin (active).
* Pregnancy.
* Neuropsychiatric pathologies (schizophrenia, bipolarity, cognitive alteration).
* Subjects receiving any other physiotherapy treatment in the mandibular region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Change from the Baseline in the Oral Health-Related Quality of Life (OHRQoL) | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Spanish version of Oral Health Impact Profile 5 items (OHIP-5 items).Responses are presented on a 5-point ordinal scale (0, never; 1, hardly ever; 2, occasionally; 3, fairly often; and 4, very often). Summing all responses resulted in a score ranging from a minimum of 0 to a maximum of 20. A larger score indicated more negative impacts of oral health problems.

SECONDARY OUTCOMES:
Change from the Baseline in the Fear of temporomandibular movement (kinesiophobia) | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with the Spanish version of Tampa Scale for Temporomandibular Joint Disorder, an 11-item scale. The score for each item ranges from 0 (totally disagree) to 4 (totally agree), the higher the score, the greater the degree of kinesiophobia. The optimal cut-off point for considering kinesiophobia is 23 points.
Change from the Baseline in pain maladaptation | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with the Spanish version of Pain Catastrophizing Scale. It is a self-administered scale of 13 items. It comprises 3 dimensions: rumination; magnification and despair. Each item is valued from 0 to 4, with the maximum score being 52 points. The higher the score, the higher degree of catastrophizing.
Change from the Baseline in symptoms related to central sensitization | Baseline, 4 weeks after the end of the intervention at month 6, at month 12.
  Assessed with the Spanish version of Central Sensitization Inventory. It is divided in 2 parts. Part A contains a list of 25 items about how often the person experiences each symptom ("never, rarely, sometimes, often, or always"). Individual items are scored from "0" (never) to "4" (always), resulting in a total score range for all 25 items from "0" to "100." Part B is about if the person has been previously diagnosed with seven common central sensitization diagnoses (tension headaches/migraines, fibromyalgia, irritable bowel syndrome, restless leg syndrome, temporomandibular joint disorder, chronic fatigue syndrome, and multiple chemical sensitivities) and three central sensitization-related diagnoses (depression, anxiety/panic attacks, and neck injury). This part is for information only and is not scored. A score of 40 or higher has been recommended as a reasonable cutoff.
Change from the Baseline in self-efficacy expectations | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with the Spanish version of Chronic Self-efficacy Scale. It is a scale of 19 questions divided into 3 parts. The first part (8 questions) refers to whether the subject believes they are capable of carrying out different activities. The second part (6 questions) refers to whether the subject believes they are capable of carrying out a series of activities without help. The third part (5 questions) refers to the ability that the subject believes he has, at this time, to carry out a series of activities. The subject responds using an 11-point Likert-type scale (0=I do not think I am capable at all, 10=I think I am totally capable). The maximum score is 190 points. The higher the score, the higher the degree of self-efficacy.
Change from the Baseline in pain coping strategies | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with Reduced Chronic Pain Coping Strategies Questionnaire. It is a scale of 24 items. It is answered on a 5-point Likert scale (never = 1, always = 5). The first-order scales are religion (use of religious beliefs), catharsis (seeking social emotional support), distraction (avoidance by paying attention to pain), self-affirmation (not fainting, encouraging oneself), mental self-control (mental control of pain) and search for information (advice, queries about what to do). The second-order scales are called active strategies (distraction, mental self-control, self-affirmation, and information seeking) and passive strategies (religion and catharsis).
Change from the Pain intensity | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Evaluated with the numerical rating scale for pain. It's An 11-point numeric scale with 0 representing one pain extreme ("no pain") and 10 representing the other pain extreme ("pain as bad as you can imagine" and "worst pain imaginable"). The subject is asked to indicate the numeric value on the segmented scale that best describes their pain intensity. Higher scores indicate greater pain intensity. A reduction of approximately two points or a reduction of approximately 30% represented a clinically important difference.
Change from the Baseline in the functional status of the masticatory system | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with the Spanish version of Jaw Functional Limitation Scale-8 (JFLS8). A scale that evaluates 8 items on a scale from 0 (no limitation) to 10 (severe limitation). The higher the score, the greater the limitation.
Change from the Baseline in sleep difficulties | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with Athens Insomnia Scale. It is an 8-item scale. Participants are asked to score each item from 0 (no problem at all) to 3 (very serious problem). The total score ranges from 0 to 24.
Change from the Baseline in emotional state | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with the Spanish version of Hospital Anxiety and Depression Scale. 14-item questionnaire. Two subscales of 7 items each, on a 0-3 Likert scale. Odd items assess anxiety, even items assess depression, with a score range in each subscale of 0-21. Higher score, greater anxiety and depression. For both subscales, the authors suggest that scores greater than eleven would indicate "case" and greater than eight would be considered "probable case".
Change from the Baseline in oral behaviors | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with the Spanish version of Oral Behaviors Checklist. It's a self-reported questionnaire (diagnostic criteria for temporomandibular disorder, axis II assessment) used to identify and quantify the frequency of different oral habits. It is conformed by 21 questions, with each having 5 possible answers: none of the time=0; a little of the time=1; some of the time=2; most of the time=3; and all of the time=4. For the first 2 questions, which are about oral habits that occur at night, the possible answers are: none of the time=0; <1 night per month=1; 1 to 3 nights per month=2; 1 to 3 nights per week=3; and 4 to 7 nights per week=4. A score of 3 or 4 indicated that the patient had that particular oral habit.
Change from the knowledge about neurophysiology of pain and conceptualization of pain | Baseline, 4 weeks after the end of the intervention, at month 6, at month 12.
  Assessed with the Spanish version of Neurophysiology of Pain Questionnaire. It contains 12 items relating to the neurophysiology of pain. Each item has three response options: true, false, undecided. It is scored out of 12 with 1 point awarded for each correct response. A score of 0 is attributed to incorrect responses and those marked as undecided. The higher the score, the greater the knowledge about the neurophysiology of pain.
Treatment expectations | Pre-intervention
  Assessed with a questionnaire proposed by Puentedura et al (Development of a Clinical Prediction Rule to Identify Patients With Neck Pain Likely to Benefit From Thrust Joint Manipulation to the Cervical Spine). In this proposal, the subject is asked if he thinks that the treatment can help him. There are 5 possible responses: completely disagree, slightly disagree, neutral, somewhat agree, completely agree. The treatments they ask about are: education in the physiology of pain, jaw mobility exercises, jaw strength exercises, sleep hygiene, relaxation techniques, rest, avoiding bad oral habits, medication, surgery.
Degree of satisfaction with the intervention | 4 weeks after the end of the intervention
  Assessed with the Spanish version of Consumer Reports Effectiveness Scale (CRES-4). It consists of 4 items: a satisfaction question, a question to rate the degree of resolution of the main problem, a question about the emotional state before starting treatment and, finally, a question about the emotional state at the time of answering. To obtain the global score of the CRES-4, the results of the previous components are added together as represented by the following formula: CRES-4 = (20 x satisfaction) + (20 x problem solution) + [12.5 x (4 + current emotional state - pre-treatment emotional state)] Therefore, to interpret the CRES-4 globally, a score on a scale ranging from 0 to 300 points is considered. The higher the total score, the more effective the treatment according to the patient.
Adverse effects | 4 weeks after the end of the intervention
  Questionnaire in which you will be asked if you have had adverse effects. If so, the subject will be asked to specify what it consists of.

CONTACTS AND LOCATIONS:
Overall Officials: J. Édgar Ferrández-Gómez, Principal Investigator — Universidad de Murcia
Locations (1):
- Fibrofamur, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan NM. Secondary aldosteronism: with observations on the definition of hypokalemia. Am J Clin Pathol. 1970 Sep;54(3):316-23. doi: 10.1093/ajcp/54.3.316. No abstract available. PMID 4319208
- [Background] Salvetti G, Manfredini D, Bazzichi L, Bosco M. Clinical features of the stomatognathic involvement in fibromyalgia syndrome: a comparison with temporomandibular disorders patients. Cranio. 2007 Apr;25(2):127-33. doi: 10.1179/crn.2007.019. PMID 17508633
- [Background] Wintroub BU, Klickstein LB, Kaempfer CE, Austen KF. A human neutrophil-dependent pathway for generation of angiotensin II: purification and physicochemical characterization of the plasma protein substrate. Proc Natl Acad Sci U S A. 1981 Feb;78(2):1204-8. doi: 10.1073/pnas.78.2.1204. PMID 6785751
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Kim, Hyunjoong, and Seungwon Lee. Effects of Pain Neuroscience Education on Kinesiophobia in Patients with Chronic Pain: A Systematic Review and Meta-Analysis. Physical Therapy Rehabilitation Science. 2020 Dec; 9(4):309-317. doi:10.14474/ptrs.2020.9.4.309.
- [Background] Leake HB, Moseley GL, Stanton TR, O'Hagan ET, Heathcote LC. What do patients value learning about pain? A mixed-methods survey on the relevance of target concepts after pain science education. Pain. 2021 Oct 1;162(10):2558-2568. doi: 10.1097/j.pain.0000000000002244. PMID 33960326
- [Background] Shala R, Roussel N, Lorimer Moseley G, Osinski T, Puentedura EJ. Can we just talk our patients out of pain? Should pain neuroscience education be our only tool? J Man Manip Ther. 2021 Feb;29(1):1-3. doi: 10.1080/10669817.2021.1873259. Epub 2021 Jan 11. No abstract available. PMID 33427587
- [Background] Watson JA, Ryan CG, Cooper L, Ellington D, Whittle R, Lavender M, Dixon J, Atkinson G, Cooper K, Martin DJ. Pain Neuroscience Education for Adults With Chronic Musculoskeletal Pain: A Mixed-Methods Systematic Review and Meta-Analysis. J Pain. 2019 Oct;20(10):1140.e1-1140.e22. doi: 10.1016/j.jpain.2019.02.011. Epub 2019 Mar 1. PMID 30831273
- [Background] Siddall B, Ram A, Jones MD, Booth J, Perriman D, Summers SJ. Short-term impact of combining pain neuroscience education with exercise for chronic musculoskeletal pain: a systematic review and meta-analysis. Pain. 2022 Jan 1;163(1):e20-e30. doi: 10.1097/j.pain.0000000000002308. PMID 33863860
- [Background] Shaffer SM, Brismee JM, Courtney CA, Sizer PS. The status of temporomandibular and cervical spine education in credentialed orthopedic manual physical therapy fellowship programs: a comparison of didactic and clinical education exposure. J Man Manip Ther. 2015 Feb;23(1):51-6. doi: 10.1179/2042618614Y.0000000087. PMID 26674266
- [Background] Romm MJ, Ahn S, Fiebert I, Cahalin LP. A Meta-Analysis of Therapeutic Pain Neuroscience Education, Using Dosage and Treatment Format as Moderator Variables. Pain Pract. 2021 Mar;21(3):366-380. doi: 10.1111/papr.12962. Epub 2020 Nov 22. PMID 33131210
- [Background] Zheng T, Holford TR, Ma Z, Ward BA, Flannery J, Boyle P. Continuing increase in incidence of germ-cell testis cancer in young adults: experience from Connecticut, USA, 1935-1992. Int J Cancer. 1996 Mar 15;65(6):723-9. doi: 10.1002/(SICI)1097-0215(19960315)65:63.0.CO;2-0. PMID 8631581
- [Background] Figueiro C, Knorst JK, Fensterseifer CK, Folchini S, Milanesi JM, Bernardon Silva T, Marquezan M. Changes in oral health-related quality of life after self-care treatment in patients with myofascial pain. Cranio. 2024 Mar;42(2):199-205. doi: 10.1080/08869634.2021.1922229. Epub 2021 Apr 30. PMID 33928869
- [Background] de Freitas RF, Ferreira MA, Barbosa GA, Calderon PS. Counselling and self-management therapies for temporomandibular disorders: a systematic review. J Oral Rehabil. 2013 Nov;40(11):864-74. doi: 10.1111/joor.12098. Epub 2013 Sep 18. PMID 24102692
- [Background] Michelotti A, Iodice G, Vollaro S, Steenks MH, Farella M. Evaluation of the short-term effectiveness of education versus an occlusal splint for the treatment of myofascial pain of the jaw muscles. J Am Dent Assoc. 2012 Jan;143(1):47-53. doi: 10.14219/jada.archive.2012.0018. PMID 22207667
- [Background] Michelotti A, de Wijer A, Steenks M, Farella M. Home-exercise regimes for the management of non-specific temporomandibular disorders. J Oral Rehabil. 2005 Nov;32(11):779-85. doi: 10.1111/j.1365-2842.2005.01513.x. PMID 16202040
- [Background] Aggarwal VR, Wu J, Fox F, Howdon D, Guthrie E, Mighell A. Implementation of biopsychosocial supported self-management for chronic primary oro-facial pain including temporomandibular disorders: A theory, person and evidence-based approach. J Oral Rehabil. 2021 Oct;48(10):1118-1128. doi: 10.1111/joor.13229. Epub 2021 Jul 27. PMID 34273180
- [Background] Eliassen M, Hjortsjo C, Olsen-Bergem H, Bjornland T. Self-exercise programmes and occlusal splints in the treatment of TMD-related myalgia-Evidence-based medicine? J Oral Rehabil. 2019 Nov;46(11):1088-1094. doi: 10.1111/joor.12856. Epub 2019 Jul 21. PMID 31286551
- [Background] Michelotti A, Steenks MH, Farella M, Parisini F, Cimino R, Martina R. The additional value of a home physical therapy regimen versus patient education only for the treatment of myofascial pain of the jaw muscles: short-term results of a randomized clinical trial. J Orofac Pain. 2004 Spring;18(2):114-25. PMID 15250431
- [Background] Shimada A, Ishigaki S, Matsuka Y, Komiyama O, Torisu T, Oono Y, Sato H, Naganawa T, Mine A, Yamazaki Y, Okura K, Sakuma Y, Sasaki K. Effects of exercise therapy on painful temporomandibular disorders. J Oral Rehabil. 2019 May;46(5):475-481. doi: 10.1111/joor.12770. Epub 2019 Feb 19. PMID 30664815
- [Background] Haggman-Henrikson B, Wiesinger B, Wanman A. The effect of supervised exercise on localized TMD pain and TMD pain associated with generalized pain. Acta Odontol Scand. 2018 Jan;76(1):6-12. doi: 10.1080/00016357.2017.1373304. Epub 2017 Sep 4. PMID 28870137
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Best N, Best S, Loudovici-Krug D, Smolenski UC. Measurement of mandible movements using a vernier caliper--an evaluation of the intrasession-, intersession- and interobserver reliability. Cranio. 2013 Jul;31(3):176-80. doi: 10.1179/crn.2013.028. PMID 23971158
- [Background] Ohrbach R, Larsson P, List T. The jaw functional limitation scale: development, reliability, and validity of 8-item and 20-item versions. J Orofac Pain. 2008 Summer;22(3):219-30. PMID 18780535
- [Background] Gomes MB, Guimaraes JP, Guimaraes FC, Neves AC. Palpation and pressure pain threshold: reliability and validity in patients with temporomandibular disorders. Cranio. 2008 Jul;26(3):202-10. doi: 10.1179/crn.2008.027. PMID 18686497
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Humphrey SM, Gavin JB, Herdson PB. Catecholamine-depletion and the no-reflow phenomenon in anoxic and ischaemic rat hearts. J Mol Cell Cardiol. 1982 Mar;14(3):151-61. doi: 10.1016/0022-2828(82)90113-4. No abstract available. PMID 7108970
- [Background] John MT, Omara M, Su N, List T, Sekulic S, Haggman-Henrikson B, Visscher CM, Bekes K, Reissmann DR, Baba K, Schierz O, Theis-Mahon N, Fueki K, Stamm T, Bondemark L, Oghli I, van Wijk A, Larsson P. RECOMMENDATIONS FOR USE AND SCORING OF ORAL HEALTH IMPACT PROFILE VERSIONS. J Evid Based Dent Pract. 2022 Mar;22(1):101619. doi: 10.1016/j.jebdp.2021.101619. Epub 2021 Aug 10. PMID 35219460
- [Background] Visscher CM, Ohrbach R, van Wijk AJ, Wilkosz M, Naeije M. The Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-TMD). Pain. 2010 Sep;150(3):492-500. doi: 10.1016/j.pain.2010.06.002. Epub 2010 Jul 3. PMID 20598804
- [Background] Nelson EA, Weikert M, Phillips JA. Pediatric treatment costs and the HIV epidemic. J Trop Pediatr. 1995 Aug;41(4):250. doi: 10.1093/tropej/41.4.250. No abstract available. PMID 7563282
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Cabrera V, Martín-Aragón M, Terol M, Núñez R, Pastor M. Escala de Ansiedad y Depresión Hospitalaria (HAD) en fibromialgia: Análisis de sensibilidad y especificidad. La Terapia psicológica. 2015; 33(3): 181-193. https://dx.doi.org/10.4067/S0718-48082015000300003
- [Background] Herrero MJ, Blanch J, Peri JM, De Pablo J, Pintor L, Bulbena A. A validation study of the hospital anxiety and depression scale (HADS) in a Spanish population. Gen Hosp Psychiatry. 2003 Jul-Aug;25(4):277-83. doi: 10.1016/s0163-8343(03)00043-4. PMID 12850660
- [Background] Enomoto K, Adachi T, Yamada K, Inoue D, Nakanishi M, Nishigami T, Shibata M. Reliability and validity of the Athens Insomnia Scale in chronic pain patients. J Pain Res. 2018 Apr 16;11:793-801. doi: 10.2147/JPR.S154852. eCollection 2018. PMID 29713192
- [Background] Gomez-Benito J, Ruiz C, Guilera G. A Spanish version of the Athens Insomnia Scale. Qual Life Res. 2011 Aug;20(6):931-7. doi: 10.1007/s11136-010-9827-x. Epub 2011 Jan 6. PMID 21210225
- [Background] Puentedura EJ, Cleland JA, Landers MR, Mintken PE, Louw A, Fernandez-de-Las-Penas C. Development of a clinical prediction rule to identify patients with neck pain likely to benefit from thrust joint manipulation to the cervical spine. J Orthop Sports Phys Ther. 2012 Jul;42(7):577-92. doi: 10.2519/jospt.2012.4243. Epub 2012 May 14. PMID 22585595
- [Background] Feixas G, Pucurull O, Roca C, Paz C, García-Grau E, Bados A. Escala de satisfacción con el tratamiento recibido (CRES-4): La versión en español. Revista de Psicoterapia. 2012; 23(89): 51-58. DOI: 10.33898/rdp.v23i89.639
- [Background] Xu L, Cai B, Fan S, Lu S, Dai K. Association of Oral Behaviors with Anxiety, Depression, and Jaw Function in Patients with Temporomandibular Disorders in China: A Cross-Sectional Study. Med Sci Monit. 2021 May 17;27:e929985. doi: 10.12659/MSM.929985. PMID 33999914
- [Background] Haggman-Henrikson B, M Visscher C, Wanman A, Ljotsson B, C Peck C, Lovgren A. Even mild catastrophic thinking is related to pain intensity in individuals with painful temporomandibular disorders. J Oral Rehabil. 2021 Nov;48(11):1193-1200. doi: 10.1111/joor.13251. Epub 2021 Sep 15. PMID 34462940
- [Background] Osman A, Barrios FX, Kopper BA, Hauptmann W, Jones J, O'Neill E. Factor structure, reliability, and validity of the Pain Catastrophizing Scale. J Behav Med. 1997 Dec;20(6):589-605. doi: 10.1023/a:1025570508954. PMID 9429990
- [Background] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Background] Catley MJ, O'Connell NE, Moseley GL. How good is the neurophysiology of pain questionnaire? A Rasch analysis of psychometric properties. J Pain. 2013 Aug;14(8):818-27. doi: 10.1016/j.jpain.2013.02.008. Epub 2013 May 4. PMID 23651882
- [Background] Clinton JJ, McCormick K, Besteman J. Enhancing clinical practice. The role of practice guidelines. Am Psychol. 1994 Jan;49(1):30-3. doi: 10.1037//0003-066x.49.1.30. PMID 8122815
- [Background] Neblett R, Hartzell MM, Cohen H, Mayer TG, Williams M, Choi Y, Gatchel RJ. Ability of the central sensitization inventory to identify central sensitivity syndromes in an outpatient chronic pain sample. Clin J Pain. 2015 Apr;31(4):323-32. doi: 10.1097/AJP.0000000000000113. PMID 24806467
- [Background] Neblett R, Hartzell MM, Mayer TG, Cohen H, Gatchel RJ. Establishing Clinically Relevant Severity Levels for the Central Sensitization Inventory. Pain Pract. 2017 Feb;17(2):166-175. doi: 10.1111/papr.12440. Epub 2016 Mar 15. PMID 26989894
- [Background] Scerbo T, Colasurdo J, Dunn S, Unger J, Nijs J, Cook C. Measurement Properties of the Central Sensitization Inventory: A Systematic Review. Pain Pract. 2018 Apr;18(4):544-554. doi: 10.1111/papr.12636. Epub 2017 Nov 20. PMID 28851012
- [Background] Cuesta-Vargas AI, Roldan-Jimenez C, Neblett R, Gatchel RJ. Cross-cultural adaptation and validity of the Spanish central sensitization inventory. Springerplus. 2016 Oct 21;5(1):1837. doi: 10.1186/s40064-016-3515-4. eCollection 2016. PMID 27818875
- [Background] Martín-Aragón M, Pastor M.A, Rodríguez-Marín J, Marcha M.J, Lledó A, López-Roig. Percepción de autoeficacia en dolor crónico. Adaptación y validación de la Chronic Pain Self-efficacy Scale. Revista de Psicología de la Salud. 1999;11(1):51-76. DOI: https://doi.org/10.21134/pssa.v11i1.799
- [Background] Pastor J, Monsalve V. Validation of the reduced chronic pain coping questionnaire (CAD-R). Revista de la Sociedad Española del Dolor. 1 de octubre de 2004;11(7):407-14.
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273
- [Background] Lindfors E, Magnusson T, Ernberg M. Effect of Therapeutic Jaw Exercises in the Treatment of Masticatory Myofascial Pain: A Randomized Controlled Study. J Oral Facial Pain Headache. 2020 Fall;34(4):364-373. doi: 10.11607/ofph.2670. PMID 33290442
- [Background] Brain K, Burrows TL, Rollo ME, Chai LK, Clarke ED, Hayes C, Hodson FJ, Collins CE. A systematic review and meta-analysis of nutrition interventions for chronic noncancer pain. J Hum Nutr Diet. 2019 Apr;32(2):198-225. doi: 10.1111/jhn.12601. Epub 2018 Oct 7. PMID 30294938
- [Background] Stepanski EJ, Wyatt JK. Use of sleep hygiene in the treatment of insomnia. Sleep Med Rev. 2003 Jun;7(3):215-25. doi: 10.1053/smrv.2001.0246. PMID 12927121
- [Background] Nijs J, Roose E, Lahousse A, Mostaqim K, Reynebeau I, De Couck M, Beckwee D, Huysmans E, Bults R, van Wilgen P, Leysen L. Pain and Opioid Use in Cancer Survivors: A Practical Guide to Account for Perceived Injustice. Pain Physician. 2021 Aug;24(5):309-317. PMID 34323432
- [Background] do-Nascimento R, Maia J, de-Medeiros S, Silva HJ, Lins C, Souza MC. Pain education to women with fibromyalgia using the DolorÔmetro game. Brazilian Journal Of Pain. 2020; 3(2): 131-135. http://dx.doi.org/10.5935/2595-0118.20200026
- [Background] Vlasova EB. [The significance of the means of administering a reacting dose of toxin for determining the level of immunity in mice immunized with type A C1. oedematiens toxoid]. Zh Mikrobiol Epidemiol Immunobiol. 1974 Aug;(8):132-3. No abstract available. Russian. PMID 4450869
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728